CLINICAL TRIAL: NCT01179607
Title: A Randomized, Double Blind, Placebo Controlled, Phase II, Dose-titration Trial to Explore the Safety, Tolerability, Pharmacokinetic Profile and Efficacy of M0002 in Cirrhotic Subjects With Ascites and Hypo- or Normonatraemia.
Brief Title: Study of Efficacy of a Vasopressin 2 Receptor Antagonist M0002 for Treatment of Ascites in Cirrhotic Subjects With Hypo- or Normonatraemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Movetis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M0002-BEL-C201
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-07

CONDITIONS: Cirrhotic Ascites

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- M0002 (Active Comparator): * Started at 0.3 mg/day and increased every 3 days (to 1, 3 and 6 mg/day)
  * for hyponatraemic subjects: dose was increased until the evening serum level was between 132 mmol/l and 145 mmol/l;
  * for normonatraemic subjects the dose was increased until a 500 ml increase in the 24-h urine volume compared with Day-1 was reached.
  Once the required response or max dose was achieved, subjects entered a maintenance phase where they remained on the same dose of M0002 or placebo until 15 days.
  Interventions: Drug: M0002
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M0002
  Arms: M0002
Drug: Placebo
  Arms: Placebo

SUMMARY:
M0002, an orally active, selective non-peptidergic antagonist of the vasopressin V2 receptor inhibits vasopressin-induced water reabsorption from the kidney. Therefore the aquaretic effect of M0002 has a potential clinical benefit in the treatment of ascites and hyponatreamia in cirrhotic patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subjects with any form of cirrhosis with ascites and who had at least 1 paracentesis of at least 4 liter in the last 6 months.
2. Dose of diuretics of spironolactone and furosemide was to be stable for at least one week prior to the screening visit or subject was refractory to diuretics.
3. Subjects had to have been on a salt restricted diet (< 5.2 grams sodium/day, 90 mmol) during the screening period prior to the trial drug administration.
4. Other treatment for the management of cirrhosis and ascites should be stable for at least 2 weeks prior to trial drug administration.
5. Child-Pugh B and C liver cirrhosis score lower than 12.
6. Subjects with hyponatraemia with sodium level between 120 and 132 mmol/l or normonatraemia with sodium level between 133 and 145 mmol/l measured at screening visit and day 1.

Main Exclusion Criteria:

1. Women of child bearing potential (WOCBP)
2. Functional transjugular intrahepatic portasystemic stent shunt (TIPS), peritoneovenous shunt
3. Liver transplantation
4. Budd-Chiari syndrome
5. Unstable hepatic disease (acute hepatitis, AST or ALT > 5 x upper limit of normal, bilirubin > 10 mg/dL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Plasma sodium levels, weight, number of paracentesis | 15 days